CLINICAL TRIAL: NCT02295787
Title: Intranasal Ketamine for Late-Life Depression and Suicidal Ideation
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No funding
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Dawn F Ionescu, Assistant in Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014D006212
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Depression; Suicide; Suicidal Ideation
Keywords: Depression; Suicide; Suicidal Ideation; Ketamine; Late-Life
MeSH Terms: conditions — Depression; Suicide; Suicidal Ideation | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine (Experimental): Intranasal Ketamine 50mg administered six times over three weeks.
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): Intranasal saline solution administered six times over three weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — Intranasal ketamine for late-life depression and suicidal ideation.
  Arms: Ketamine
Drug: Placebo
  Arms: Placebo

SUMMARY:
The investigators of this study plan to investigate the feasibility and efficacy of repeated doses of intranasal ketamine in severely depressed patients who are at least 65 years of age and experiencing suicidal ideation. The results of the study could lead to development of new strategies for treating depression.

ELIGIBILITY:
Inclusion Criteria:

1) be ≥65 years old, 2) provide written informed consent, 3) meet criteria for a primary psychiatric diagnosis of major depressive disorder according to the Structured Clinical Interview for DSM-IV (SCID) and have a HDRS28 total score ≥20; depression may have started at any time point in their life, and certain co-morbid diagnoses (e.g., anxiety disorders) will be allowed insofar as they are not the primary psychiatric diagnosis, 4) have a history of ≥2 failed medication trials during the current episode (per the Massachusetts General Hospital Antidepressant Treatment History Questionnaire; MGH ATRQ), 5) endorse suicidal ideation for more than 2 months, per the Columbia Suicide Severity Rating Scale (C-SSRS) and have a HDRS28 suicide item score ≥1 (thoughts that life isn't worth living), 6) be on a stable antidepressant regimen for ≥14 days prior to Study Phase II, 7) maintain a treating psychiatrist who is in agreement with study participation, and 8) have a reliable chaperone accompany them home following the completion of the intranasal administration.

Exclusion Criteria:

* Patients will be excluded if any of the following criteria are met: 1) Delirium or dementia diagnosis, 2) unstable medical illness, 3) history of clinically significant cardiovascular disease or electrocardiogram (EKG) findings, or medical conditions that put the patient at risk for possible cardiac side effects, 4) history of multiple adverse drug reactions, 5) current/past history of psychotic disorders or homicidality, 6) active substance use disorders (except nicotine and caffeine) within the past six months, positive urine toxicology screen, or past history of ketamine abuse, 7) requirement of excluded medications (narcotics, barbiturates, theophylline, or St. John's Wort), or 8) concurrent or recent participation in other research studies.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS) | Up to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Dawn F Ionescu, MD, Principal Investigator — Massachusetts General Hospital